CLINICAL TRIAL: NCT03528239
Title: The Use of Hospital Outpatient Clinics and Emergency Department by Refugee Patients in Turkey
Brief Title: The Use of Hospital and Emergency Department of Refugee Patients
Status: Completed | Type: Observational
Sponsor: Nevsehir Public Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Nevşehir
Record Dates: First submitted 2018-04-30; First posted 2018-05-17 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Refugees; Health Care; Outpatients; Emergency Departments
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Refugee patients — To investigate characteristics of outpatient visits of refugee patients

SUMMARY:
After Middle Eastern crisis, millions people were forced to migrate to European countries and especially neighboring countries. In Turkey, cities which are closed to east of border, face to cope more refugees' health care than those of other cities. The incidence of admission of hospital outpatient clinics and emergency department by refugee patients is not known clearly in our city, Nevsehir. In this study, we wanted to investigate use of health care among these patients in Nevsehir in Turkey.

ELIGIBILITY:
Inclusion Criteria:

All patients who visited an outpatient clinic and emergency department.

Exclusion Criteria:

Patients who have missing records.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Refugee patients are registered in the hospital system in a different way than that of others. We will use these datas as recorded refugees. And also, we will use the number of other visits to calculate the incidence of visits of refugees.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
The incidence of outpatient clinics and emergency department use by refugee patients | 2014-2017
  Hospital outpatient clinics and emergency department use by refugee patients in a secondary care hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Nevsehir State Hospital, Nevşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes